CLINICAL TRIAL: NCT07086729
Title: Development of a CT-Derived Risk Score to Guide Treatment Decision: Tracheal Stenosis Morphology and Attenuation Score (TSMAS)
Brief Title: CT-Based Scoring System to Predict Surgical Need in Tracheal Stenosis (TSMAS Study)
Status: Not yet recruiting | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Caner İşevi, MD, Principal Investigator, Ondokuz Mayıs University
Other Study IDs: B.30.2.ODM.0.20.08/ 457
Record Dates: First submitted 2025-07-10; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Tracheal Stenosis
Keywords: Tracheal Stenosis; Postintubation Stenosis; Hounsfield Unit; Morphologic Scoring; Computed Tomography
MeSH Terms: conditions — Tracheal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tracheal Stenosis Patients: Patients diagnosed with tracheal stenosis whose thoracic CT scans were retrospectively analyzed to evaluate morphological and densitometric parameters. No intervention was applied; data were used to develop a CT-based risk score (TSMAS) to predict the need for surgical treatment.
  Interventions: Other: CT-Based Morphologic and Attenuation Scoring

INTERVENTIONS:
Other: CT-Based Morphologic and Attenuation Scoring — Retrospective analysis of CT images to extract morphological and Hounsfield Unit (HU) parameters for development of a predictive scoring model (TSMAS). No clinical or therapeutic intervention was performed.

SUMMARY:
This study aims to develop a CT-based scoring system to help predict whether patients with tracheal stenosis will require surgical treatment or can be managed with endoscopic procedures. Using retrospective data, researchers will evaluate CT scans of patients diagnosed with tracheal stenosis to measure features such as airway diameter, wall thickness, and tissue density (measured in Hounsfield Units). The goal is to create a non-invasive, reproducible, and objective tool-called the Tracheal Stenosis Morphology and Attenuation Score (TSMAS)-that can support clinical decision-making and improve treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosed with tracheal stenosis
* Underwent thoracic CT imaging at the time of diagnosis
* CT scans available in adequate quality and in DICOM format
* No prior surgical treatment for tracheal stenosis before CT imaging

Exclusion Criteria:

* Tracheal stenosis due to malignancy, foreign body, or tracheobronchial tumors
* History of tracheal surgery before CT imaging
* Poor quality CT images (e.g., motion artifacts, incomplete tracheal segments)
* Patients with a history of radiotherapy (RT) to the neck or mediastinum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (aged 18 and older) diagnosed with tracheal stenosis, who underwent thoracic CT imaging at the time of diagnosis. All patients were treated or followed at Ondokuz Mayıs University Hospital between 2000 and 2025. Only patients with sufficient-quality DICOM-format CT scans and no prior tracheal surgery or radiotherapy were included.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Prediction of Surgical Requirement Based on Tracheal Diameter on Initial CT | From initial diagnosis to surgical decision (up to 12 months)
  Evaluation of whether smaller tracheal diameter on initial CT is associated with need for surgery.
  Unit of Measure: millimeters
Prediction of Surgical Requirement Based on Tracheal Wall Thickness on Initial CT | From initial diagnosis to surgical decision (up to 12 months)
  Evaluation of whether increased tracheal wall thickness on initial CT predicts surgical need.
  Unit of Measure: millimeters
Prediction of Surgical Requirement Based on HU Values of the Stenotic Segment on CT | From initial diagnosis to surgical decision (up to 12 months)
  Evaluation of whether high HU values in the stenotic segment predict surgical need.
  Unit of Measure: Hounsfield Units (HU)

IPD SHARING:
Plan to Share IPD: Yes